CLINICAL TRIAL: NCT01400529
Title: Etude 3000 ARTHROSES Symptomatic Knee and Hip Osteoarthritis Prevalence Survey. Programme de Recherche du Groupe Qualité de Vie, de la Section Epidémiologie et de la Section Arthrose de la Société Française de Rhumatologie
Brief Title: Etude 3000 ARTHROSES Symptomatic Knee and Hip Osteoarthritis Prevalence Survey
Acronym: 3000ARTHROSE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Philippe Boulangé, direction de la recherche et de l'innovation, Central Hospital, Nancy, France
Other Study IDs: 906297
Record Dates: First submitted 2007-07-05; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2007-07

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; knee; hip; population based
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Nationwide descriptive epidemiology survey aiming to determine lower limb OA prevalence, based on a validated method previously used to assess inflammatory rheumatism (rheumatoid arthritis and spondylarthropathy) prevalence in France.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative disease progressively affecting joint cartilage and subchondral bone, leading to pain, limited range of motion and functional impairment. Knee and hip are the more frequently affected joints. There is no treatment able to cure OA or at least to slow down cartilage damage. Thus, when symptomatic treatments become ineffective, joint prosthetic replacement is the unique solution.

There is a substantial lack of information about osteoarthritis (OA) epidemiology in France, as well as in other European countries, which becomes more and more critical with population aging. The need for additional knowledge was outlined in the law about public health priorities in France, published on August 9th, 2004. In this document, a specific call is made for additional investigation on functional limitations, disability and quality of life modification of people affected by OA.

Up to now, available information is mainly limited to short- or medium-term studies, conducted in clinic-based samples. Thus, based on demography and public health conclusions, implementing population-based epidemiologic studies is required in order to improve scientific knowledge with regards to :

* prevalence of symptomatic OA,
* its natural history over years and potential prognostic factors influencing the disease,
* its impact in terms of quality of life changes, disability, lack of autonomy and health resource use.

Our expert group, which has a substantial experience in osteoarthritis, epidemiology and health service research, has developed a 2-part research program aiming to help answering to OA-related public health questions:

* Part 1: a nationwide descriptive epidemiology survey aiming to determine lower limb OA prevalence, based on a validated method previously used to assess inflammatory rheumatism (rheumatoid arthritis and spondylarthropathy) prevalence in France.
* Part 2: the constitution of a population-based cohort of OA patients, aiming to collect clinical, biologic and radiological data about OA natural history, predictors of structural progression, consequences on quality of life, function and health resource use.

The present study is the part 1 of the program

ELIGIBILITY:
Inclusion Criteria:

* age 40-75
* adults in households representative of the French population for age, sex, area of living and number of household members.

Exclusion Criteria:

Ages: 40 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: population based
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2007-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Guillemin, MD, PhD, Principal Investigator — Societe Francaise de Rhumatologie
Locations (6):
- France (6):
  - Service de Rhumatologie. CHU d'Amiens, Amiens
  - Service de Rhumatologie. CHU de la Cavale Blanche, Brest
  - Centre d'Epidémiologie Clinique. Service de rhumatologie. CHU Nancy, Nancy
  - Service de Rhumatologie. CHU L'Archet 1, Nice
  - Service de Rhumatologie. Hôpital de la Pitié-Salpêtrière, Paris
  - Service de Rhumatologie. Hôpital Rangueil, Toulouse

REFERENCES:
- [Derived] Guillemin F, Rat AC, Mazieres B, Pouchot J, Fautrel B, Euller-Ziegler L, Fardellone P, Morvan J, Roux CH, Verrouil E, Saraux A, Coste J; 3000 Osteoarthritis group. Prevalence of symptomatic hip and knee osteoarthritis: a two-phase population-based survey. Osteoarthritis Cartilage. 2011 Nov;19(11):1314-22. doi: 10.1016/j.joca.2011.08.004. Epub 2011 Aug 16. PMID 21875676